CLINICAL TRIAL: NCT03087175
Title: Impact of Polyethylene Terephthalate Micronet Mesh-Covered Stent (MGuard) on Coronary Microcirculation's Lesions in Patients With ST or Non ST-segment Elevation Myocardial Infarction (STE and NSTE-ACS): Assessment by Index of Microcirculatory Resistance (IMR)
Brief Title: MGuard Stent and Microcirculation
Acronym: GUARDIANCORY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC15.311
Record Dates: First submitted 2016-11-14; First posted 2017-03-22 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Atherosclerosis; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Cardiovascular Diseases | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MGuard stent (Experimental): MGuard stent is a novel thin-strut metal stent with a polyethylene terephthalate micronet covering designed to trap and exclude thrombus and friable atheromatous debris to prevent distal embolization
  Interventions: Device: MGuard stent
- Drug eluting stent and bare metal stent (Active Comparator): Drug eluting stent and bare metal stent
  Interventions: Device: Drug eluting stent and bare metal stent

INTERVENTIONS:
Device: MGuard stent — MGuard micronet mesh-covered stent in treatment of STE and NSTE-ACS
  Other Names: MGuard micronet mesh-covered stent
  Arms: MGuard stent
Device: Drug eluting stent and bare metal stent — Drug eluting stent and bare metal stent in treatment of STE and NSTE-ACS For example, Resolute Onyx
  Other Names: Resolute Onyx
  Arms: Drug eluting stent and bare metal stent

SUMMARY:
NSTE-ACS represents the most frequent indication for coronary angiography and percutaneous coronary intervention (PCI) worldwide. PCI permit to reestablished coronary flow but effectiveness of PCI within thrombus containing lesions is limited by the risk of occurrence of distal embolization and no-reflow phenomenon. Distal embolization lead to coronary microcirculation lesions. This complication is related to poor prognosis.

MGuard stent is a stainless-steel closed cell stent covered with an ultra-thin polymer mesh sleeve, which allows to prevent distal embolization during percutaneous coronary intervention in ST-segment-elevation myocardial infarction.

Index of microcirculatory resistance (IMR) is a validated method to assess coronary microcirculation.

Accordingly, the purpose of this study is to demonstrate that MGuard micronet mesh-covered stent prevent distal embolization and microvascular reperfusion impairment during primary PCI, compared with a bare metal stent (BMS) and drug eluting stent (DES) in patients with NSTE-ACS, assessed by Index of microcirculatory resistance.

DETAILED DESCRIPTION:
GUARDIANCORY study is a multicentre, prospective, randomized, non inferiority, open-label trial with a planned inclusion of 52 patients with STE and NSTE ACS and prescribed PCI. Patients will be randomized to benefiting either DES /BMS implantation (n=26) or MGuard stent (n=26) on the culprit lesion. Assessment of coronary microcirculation will be done by IMR immediately after PCI by using a pressure-temperature sensor-tipped coronary wire, thermodilution-derived.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients affiliated to social security
* Patients with an NSTEMI or STEMI (1)
* Thrombus containing coronary lesions on angiography (TIMI thrombus grade ≥ 3)
* Eligible patients for revascularization with angioplasty
* Patients consenting to participate in the study.

Exclusion Criteria:

* Age < 18 years
* Prior myocardial infarction
* Prior CABG
* Inability to comply with the protocol
* Major patient protected by law (article L1121-8),
* Person deprived of liberty (article L1121-8),
* Pregnant woman
* Breastfeeding women
* Patient with terminal illness,
* Terminal Renal failure
* Allergy to iodine
* Adenosine's contraindications: Asthmatic patients, Second- or third-degree AV block without a pacemaker or sick sinus syndrome. Systolic blood pressure less than 90mmHg. Recent use of dipyridamole or dipyridamole-containing medications, Methyl xanthenes such as aminophylline caffeine or theobromine block the effect of adenosine and should be held for at least 12 hours prior to the test. Known hypersensitivity to adenosine. Unstable acute myocardial infarction or acute coronary syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12; Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Index of microcirculatory resistance (IMR) | During the 2 hours after randomization
  Index of microcirculatory resistance (IMR) will be measured with a pressure sensor/thermistor-tipped guidewire

SECONDARY OUTCOMES:
TIMI flux on angiography | During the 2 hours after randomization
Grade blush on angiography | During the 2 hours after randomization
TIMI frame count measure | During the 2 hours after randomization
Measure of risk area by BARI-Score | During the 2 hours after randomisation
ST-segment resolution defined by >70% ST-segment resolution on EKG post angioplasty compared to initial EKG | During the 24 hours after randomization
Enzymatic cycle with measure of troponin T and CPK pick | 7 days after randomization
Measure of wall motion score (WMS) by echocardiography | 2, 7 days after randomization, 6 month follow-up
Measure of 2D strain by echocardiography | 2, 7 days after randomization, 6 month follow-up
Cardiological follow up to detect intrastent restenosis | 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BARONE-ROCHETTE, MD, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (2):
- France (2):
  - Annecy Hospital, Annecy
  - University Hospital Grenoble, Grenoble

REFERENCES:
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Silen W, Machen TE, Forte JG. Acid-base balance in amphibian gastric mucosa. Am J Physiol. 1975 Sep;229(3):721-30. doi: 10.1152/ajplegacy.1975.229.3.721. PMID 2015
- [Background] Pride YB, Mohanavelu S, Zorkun C, Kunadian V, Giugliano RP, Newby LK, Braunwald E, Califf RM, Harrington RA, Gibson CM; EARLY ACS Investigators. Association between angiographic complications and clinical outcomes among patients with acute coronary syndrome undergoing percutaneous coronary intervention: an EARLY ACS (Early Glycoprotein IIb/IIIa Inhibition in Non-ST-Segment Elevation Acute Coronary Syndrome) angiographic substudy. JACC Cardiovasc Interv. 2012 Sep;5(9):927-35. doi: 10.1016/j.jcin.2012.05.007. PMID 22995880
- [Background] Gibson CM, Kirtane AJ, Morrow DA, Palabrica TM, Murphy SA, Stone PH, Scirica BM, Jennings LK, Herrmann HC, Cohen DJ, McCabe CH, Braunwald E; TIMI Study Group. Association between thrombolysis in myocardial infarction myocardial perfusion grade, biomarkers, and clinical outcomes among patients with moderate- to high-risk acute coronary syndromes: observations from the randomized trial to evaluate the relative PROTECTion against post-PCI microvascular dysfunction and post-PCI ischemia among antiplatelet and antithrombotic agents-Thrombolysis In Myocardial Infarction 30 (PROTECT-TIMI 30). Am Heart J. 2006 Oct;152(4):756-61. doi: 10.1016/j.ahj.2006.04.016. PMID 16996854
- [Background] Gibson CM, de Lemos JA, Murphy SA, Marble SJ, McCabe CH, Cannon CP, Antman EM, Braunwald E; TIMI Study Group. Combination therapy with abciximab reduces angiographically evident thrombus in acute myocardial infarction: a TIMI 14 substudy. Circulation. 2001 May 29;103(21):2550-4. doi: 10.1161/01.cir.103.21.2550. PMID 11382722
- [Background] De Bruyne B, Pijls NH, Smith L, Wievegg M, Heyndrickx GR. Coronary thermodilution to assess flow reserve: experimental validation. Circulation. 2001 Oct 23;104(17):2003-6. doi: 10.1161/hc4201.099223. PMID 11673336
- [Background] Steg PG, Dabbous OH, Feldman LJ, Cohen-Solal A, Aumont MC, Lopez-Sendon J, Budaj A, Goldberg RJ, Klein W, Anderson FA Jr; Global Registry of Acute Coronary Events Investigators. Determinants and prognostic impact of heart failure complicating acute coronary syndromes: observations from the Global Registry of Acute Coronary Events (GRACE). Circulation. 2004 Feb 3;109(4):494-9. doi: 10.1161/01.CIR.0000109691.16944.DA. Epub 2004 Jan 26. PMID 14744970
- [Background] Cuisset T, Hamilos M, Melikian N, Wyffels E, Sarma J, Sarno G, Barbato E, Bartunek J, Wijns W, De Bruyne B. Direct stenting for stable angina pectoris is associated with reduced periprocedural microcirculatory injury compared with stenting after pre-dilation. J Am Coll Cardiol. 2008 Mar 18;51(11):1060-5. doi: 10.1016/j.jacc.2007.11.059. PMID 18342222
- [Background] Holm J, Haggendal E, Lundberg D, Schersten T, Stenberg K, Wetterqvist H. Effect of lumbar sympathetic blockade and chlorpromazine-induced adrenergic alpha-receptor blockade on skin temperature in peripheral arterial diseases. J Cardiovasc Surg (Torino). 1976 Jan-Feb;17(1):69-71. PMID 1398
- [Background] Aarnoudse W, Fearon WF, Manoharan G, Geven M, van de Vosse F, Rutten M, De Bruyne B, Pijls NH. Epicardial stenosis severity does not affect minimal microcirculatory resistance. Circulation. 2004 Oct 12;110(15):2137-42. doi: 10.1161/01.CIR.0000143893.18451.0E. Epub 2004 Oct 4. PMID 15466646
- [Background] Nijveldt R, Beek AM, Hirsch A, Stoel MG, Hofman MB, Umans VA, Algra PR, Twisk JW, van Rossum AC. Functional recovery after acute myocardial infarction: comparison between angiography, electrocardiography, and cardiovascular magnetic resonance measures of microvascular injury. J Am Coll Cardiol. 2008 Jul 15;52(3):181-9. doi: 10.1016/j.jacc.2008.04.006. PMID 18617066
- [Background] Henriques JP, Zijlstra F, Ottervanger JP, de Boer MJ, van 't Hof AW, Hoorntje JC, Suryapranata H. Incidence and clinical significance of distal embolization during primary angioplasty for acute myocardial infarction. Eur Heart J. 2002 Jul;23(14):1112-7. doi: 10.1053/euhj.2001.3035. PMID 12090749
- [Background] Kaul P, Ezekowitz JA, Armstrong PW, Leung BK, Savu A, Welsh RC, Quan H, Knudtson ML, McAlister FA. Incidence of heart failure and mortality after acute coronary syndromes. Am Heart J. 2013 Mar;165(3):379-85.e2. doi: 10.1016/j.ahj.2012.12.005. Epub 2013 Jan 22. PMID 23453107
- [Background] Ng MK, Yeung AC, Fearon WF. Invasive assessment of the coronary microcirculation: superior reproducibility and less hemodynamic dependence of index of microcirculatory resistance compared with coronary flow reserve. Circulation. 2006 May 2;113(17):2054-61. doi: 10.1161/CIRCULATIONAHA.105.603522. Epub 2006 Apr 24. PMID 16636168
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] Akdeniz C, Umman S, Nisanci Y, Umman B, Bugra Z, Aslanger EK, Kaplan A, Yilmaz A, Teker E, Guz G, Polat N, Sezer M. Percutaneous coronary intervention increases microvascular resistance in patients with non-ST-elevation acute coronary syndrome. EuroIntervention. 2013 Jun 22;9(2):228-34. doi: 10.4244/EIJV9I2A38. PMID 23410633
- [Background] Fearon WF, Shah M, Ng M, Brinton T, Wilson A, Tremmel JA, Schnittger I, Lee DP, Vagelos RH, Fitzgerald PJ, Yock PG, Yeung AC. Predictive value of the index of microcirculatory resistance in patients with ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2008 Feb 5;51(5):560-5. doi: 10.1016/j.jacc.2007.08.062. PMID 18237685
- [Background] Napodano M, Ramondo A, Tarantini G, Peluso D, Compagno S, Fraccaro C, Frigo AC, Razzolini R, Iliceto S. Predictors and time-related impact of distal embolization during primary angioplasty. Eur Heart J. 2009 Feb;30(3):305-13. doi: 10.1093/eurheartj/ehn594. Epub 2009 Jan 19. PMID 19153179
- [Background] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, Ho MY, Kim HS, Loh JP, Oldroyd KG. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41. doi: 10.1161/CIRCULATIONAHA.112.000298. Epub 2013 May 16. PMID 23681066
- [Background] Stone GW, Abizaid A, Silber S, Dizon JM, Merkely B, Costa RA, Kornowski R, Abizaid A, Wojdyla R, Maehara A, Dressler O, Brener SJ, Bar E, Dudek D. Prospective, Randomized, Multicenter Evaluation of a Polyethylene Terephthalate Micronet Mesh-Covered Stent (MGuard) in ST-Segment Elevation Myocardial Infarction: The MASTER Trial. J Am Coll Cardiol. 2012 Nov 6;60(19):1975-84. doi: 10.1016/j.jacc.2012.09.004. PMID 23103033
- [Background] Jolly SS, Cairns JA, Yusuf S, Meeks B, Pogue J, Rokoss MJ, Kedev S, Thabane L, Stankovic G, Moreno R, Gershlick A, Chowdhary S, Lavi S, Niemela K, Steg PG, Bernat I, Xu Y, Cantor WJ, Overgaard CB, Naber CK, Cheema AN, Welsh RC, Bertrand OF, Avezum A, Bhindi R, Pancholy S, Rao SV, Natarajan MK, ten Berg JM, Shestakovska O, Gao P, Widimsky P, Dzavik V; TOTAL Investigators. Randomized trial of primary PCI with or without routine manual thrombectomy. N Engl J Med. 2015 Apr 9;372(15):1389-98. doi: 10.1056/NEJMoa1415098. Epub 2015 Mar 16. PMID 25853743
- [Background] Napodano M, Dariol G, Al Mamary AH, Marra MP, Tarantini G, D'Amico G, Frigo AC, Buja P, Razzolini R, Iliceto S. Thrombus burden and myocardial damage during primary percutaneous coronary intervention. Am J Cardiol. 2014 May 1;113(9):1449-56. doi: 10.1016/j.amjcard.2014.01.423. Epub 2014 Feb 12. PMID 24630783
- [Background] Layland J, Carrick D, McEntegart M, Ahmed N, Payne A, McClure J, Sood A, McGeoch R, MacIsaac A, Whitbourn R, Wilson A, Oldroyd K, Berry C. Vasodilatory capacity of the coronary microcirculation is preserved in selected patients with non-ST-segment-elevation myocardial infarction. Circ Cardiovasc Interv. 2013 Jun;6(3):231-6. doi: 10.1161/CIRCINTERVENTIONS.112.000180. Epub 2013 Jun 11. PMID 23756697